CLINICAL TRIAL: NCT03181594
Title: Clinical Evaluation of Safety and Efficacy for the ClariFix™ Cryotherapy Device in Subjects With Chronic Rhinitis
Brief Title: Evaluation of the ClariFix™ Cryotherapy Device in Subjects With Chronic Rhinitis
Acronym: FROST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arrinex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-0003
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Results first posted 2019-11-04 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-02

CONDITIONS: Chronic Rhinitis
Keywords: Cryotherapy; Cryoablation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment with the ClariFix Device (Experimental): Bilateral ablation of nasal tissue for treatment of chronic rhinitis
  Interventions: Device: ClariFix Device

INTERVENTIONS:
Device: ClariFix Device — Cryoablation in the nasal passageway using the ClariFix Device

SUMMARY:
A multi-center, prospective, non-randomized, interventional clinical trial to assess the safety and effectiveness of the ClariFix™ device when used to ablate unwanted tissue in the nose of subjects with chronic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is >21 years of age
2. Subject has moderate to severe symptoms of rhinorrhea (individual symptom rating of 2 or 3), mild to severe symptoms of congestion (individual symptom rating of 1, 2 or 3) and a minimum TNSS score of 4 (out of 12) at the time of the treatment visit, which have been present for > 6 months.
3. Subject has had documented allergy test within the last 10 years that defines whether or not subject has allergies to perennial and seasonal allergens or is willing to have one performed prior to study exit.
4. Subject has been dissatisfied with medical management, defined as usage of intranasal steroids for a minimum of 4 weeks without adequate symptom relief by the subject's assessment.
5. Subject has signed IRB-approved informed consent form

Exclusion Criteria:

1. Subject has clinically significant anatomic obstructions that in the investigator's opinion limit access to the posterior nose, including but not limited to septal deviation or perforation, nasal polyps, sinonasal tumor.
2. Subject has had any prior sinus or nasal surgery that significantly alters the anatomy of the posterior nose.
3. Subject has active nasal or sinus infection.
4. Subject has moderate to severe ocular symptoms.
5. Subject has a history of nosebleeds in the past 3 months.
6. Subject has a history of rhinitis medicamentosa.
7. Subject has had prior head or neck irradiation
8. Subject has active coagulation disorder or is receiving anti-coagulants which cannot be safely stopped for 4 weeks (excluding aspirin).
9. Subject is pregnant.
10. Subject is participating in another clinical research study.
11. Subject has an allergy or intolerance to anesthetic agent.
12. Subject has cryoglobulinemia, paroxysmal cold hemoglobinuria, cold urticaria, Raynaud's disease, and/or, open and/or infected wounds at or near the target tissue.
13. Any physical condition that in the investigator's opinion would prevent adequate study participation or pose increased risk.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2020-04-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - California Sleep Institute, East Palo Alto, California
  - Sacramento Ear, Nose, and Throat, Sacramento, California
  - San Francisco Otolaryngology Medical Group, San Francisco, California
  - Ear, Nose, and Throat Associates of South Florida, Boca Raton, Florida
  - Bethlehem Ear, Nose, and Throat, Bethlehem, Pennsylvania
  - EVMS Otolaryngology, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chang MT, Song S, Hwang PH. Cryosurgical ablation for treatment of rhinitis: A prospective multicenter study. Laryngoscope. 2020 Aug;130(8):1877-1884. doi: 10.1002/lary.28301. Epub 2019 Sep 30. PMID 31566744
- [Result] Ow RA, O'Malley EM, Han JK, Lam KK, Yen DM. Cryosurgical Ablation for Treatment of Rhinitis: Two-Year Results of a Prospective Multicenter Study. Laryngoscope. 2021 Sep;131(9):1952-1957. doi: 10.1002/lary.29453. Epub 2021 Feb 22. PMID 33616224

RESULTS

PARTICIPANT FLOW:
Period: Initial Study Protocol (12-month FU)
Arm/Group | Treatment With the ClariFix Device
Started | 100
30-day Follow-up (1 participant missed the 30-day visit but continued in later follow-up visits.) | 99
90-day Follow-up | 98
6-month Follow-up | 98
9-month Follow-up | 95
12-month Follow-up | 91
Completed | 91
Not Completed | 9
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1
Not completed — Death | 1
Period: Long-term Extension (15-24 Month FU)
Arm/Group | Treatment With the ClariFix Device
Started | 62
15-month Follow-up (Of the 91 participants who completed the 12-month visit, 28 did not consent to the long-term follow-up and 1 participant died before the long-term follow-up started resulting in 62 participants being eligible for long-term follow-up . 6/62 participants missed the 15-month missed visit.) | 56
18-month Follow-up (5/62 participants missed the 18-month visit.) | 57
21-month Follow-up (6 participants missed the 21-month visit.) | 55
24-month Follow-up | 57
Completed | 57
Not Completed | 5
Not completed — Lost to Follow-up | 3
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment With the ClariFix Device
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 96
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 90
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 100
Rhinitis subtype [Count of Participants; unit: Participants]
  Allergic | 30
  Non-allergic | 70
Baseline rTNSS [Mean (Standard Deviation); unit: units on a scale] — The reflective Total Nasal Symptom Score (rTNSS) is a validated patient-reported outcome (PRO) used to describe symptoms of rhinitis. The assessment consists of 4 nasal symptom domains (runny nose [rhinorrhea], itchy nose, sneezing, and stuffiness [nasal congestion]). Each item is rated from 0 (absent) to 3 (severe). The 4 domains are added together to provide an overall score ranging from 0 to 12.
  units on a scale | 6.14 (1.87)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Symptom Severity
Description: Effectiveness will be assessed by the mean change in nasal symptoms using the 4-symptom rTNSS (reflective Total Nasal Symptom Score). The rTNSS is the sum of 4 individual patient-rated symptom scores for rhinorrhea, nasal congestion, nasal itching, and sneezing, each evaluated using a scale of 0=None, 1=Mild, 2=Moderate, and 3=Severe. The rTNSS has a possible score of 0-12. The reflective scores are based on the participant's evaluation of symptom severity over the preceding 24 hours. A change of 1 or more is considered the minimum clinically important difference.
Time Frame: 90 days post treatment
Population: All treated participants with 90-day follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment With the ClariFix Device
Number analyzed (Participants) | 98
score on a scale | -3.1 (2.6)
Statistical Analysis 1: Comparison: Treatment With the ClariFix Device; The null hypothesis was that the mean change from baseline for the rTNSS would be 0 (no effect). Assumptions included an alpha level of 0.5 (2-tailed), 90% power, and a standard deviation of 2.5 for the mean change from baseline. A total of 68 participants was deemed adequate to test the hypothesis; Test type: Superiority; p < 0.001, t-test, 2 sided

2. Primary Outcome: Device- and/or Procedure-related Serious Adverse Events
Description: Safety will be evaluated based on the frequency of device- and/or procedure-related serious adverse events
Time Frame: 90 days post treatment
Population: All treated participants.
Measure: Number; unit: events
Arm/Group | Treatment With the ClariFix Device
Number analyzed (Participants) | 100
events | 1

3. Secondary Outcome: Change From Baseline in the Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ)
Description: The RQLQ is a validated quality of life questionnaire that evaluates functional problems associated with rhinitis. The questionnaire assess 7 domains: activities, sleep, nose symptoms, eye symptoms, non nose/eye symptoms, practical problems, and emotional function. Each question is scores on a 7-point scale (0=not impaired at all, 6=severely impaired). A domain and total scores are based on the mean of all answered items in that domain resulting in domain or total scores ranging from 0 to 6. An average change on 0.5 or more is considered a minimal clinically important difference.
Time Frame: 90 days post treatment
Population: All treated participants with 90-day follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment With the ClariFix Device
Number analyzed (Participants) | 98
score on a scale | -1.5 (1.2)
Statistical Analysis 1: Comparison: Treatment With the ClariFix Device; Test type: Superiority; p < 0.001, t-test, 2 sided

4. Other Pre Specified Outcome: Change From Baseline in Symptom Severity
Description: Median change in nasal symptoms using the 4-symptom rTNSS (reflective Total Nasal Symptom Score). The rTNSS is the sum of 4 individual patient-rated symptom scores for rhinorrhea, nasal congestion, nasal itching, and sneezing, each evaluated using a scale of 0=None, 1=Mild, 2=Moderate, and 3=Severe. The rTNSS has a possible score of 0-12. The reflective scores are based on the participant's evaluation of symptom severity over the preceding 24 hours. A change of 1 point or more is considered the minimum clinically important difference.
Time Frame: 1, 3, 6, 9, 12, 15, 18, 21, and 24 months post procedure
Population: All participants with rTNSS scores.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Treatment With the ClariFix Device
Number analyzed (Participants) | 99
score on a scale
  1-month | -3.0 [-4.0 to -2.0]
  3-month: number analyzed (Participants) | 98
  3-month | -3.0 [-4.0 to -1.0]
  6-month: number analyzed (Participants) | 98
  6-month | -3.0 [-4.0 to -2.0]
  9-month: number analyzed (Participants) | 95
  9-month | -3.0 [-4.0 to -2.0]
  12-month: number analyzed (Participants) | 91
  12-month | -3.0 [-4.0 to -1.0]
  15-month: number analyzed (Participants) | 56
  15-month | -4.0 [-5.0 to -3.0]
  18-month: number analyzed (Participants) | 57
  18-month | -3.0 [-5.0 to -2.0]
  21-month: number analyzed (Participants) | 55
  21-month | -4.0 [-5.0 to -2.0]
  24-month: number analyzed (Participants) | 57
  24-month | -4.0 [-5.0 to -2.0]
Statistical Analysis 1: Comparison: Treatment With the ClariFix Device; Test type: Superiority; p < 0.001, Wilcoxon signed rank — p<0.001 at all time periods. p<0.05 was considered statistically significant

ADVERSE EVENTS:
Time Frame: All adverse events from procedure through 9 months post treatment.
Arm/Group | Treatment With the ClariFix Device
All-Cause Mortality (participants affected / at risk) | 4/100
Serious Adverse Events (participants affected / at risk) | 9/100
Other Adverse Events (participants affected / at risk) | 0/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With the ClariFix Device (N=100)
Foot infection (Infections and infestations) | 1 (1) — HIV-positive patient developed an infection after stepping on a piece of glass at 23 days post treatment. Not related to the study device or procedure.
Colectomy (Gastrointestinal disorders) | 1 (1) — Patient with history of colon cancer had a partial colectomy at 250 days post treatment. Not related to the study device or procedure.
Sacroiliac joint dysfunction (Musculoskeletal and connective tissue disorders) | 1 (1) — Patient underwent surgeries to treat pre-existing bilateral sacroiliac joint dysfunction at 64 and 113 days post treatment. Not related to the study device or procedure.
Retained pledget/epistaxis (Surgical and medical procedures) | 1 (2) — A retained pledget was removed from the patient's nose 19 days post treatment and resulted in profuse epistaxis. The event was related to the study procedure.
Myocardial infarction (Cardiac disorders) | 1 (1) — Myocardial infarction with stent placement at 359 days post procedure. Not related to study device or procedure.
Carotid stenosis (Vascular disorders) | 1 (1) — Carotid stenosis treated with surgery at 711 days post procedure. Not related to the study device or procedure.
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) — Participants with various cancers (breast, gastric, liver, and brain) died during the study. None of the deaths were related to the study device or procedure.
Sinus bradycardia (Cardiac disorders) | 1 (1) — Participant underwent pacemaker placement at 592 days post procedure. Not related to the study device or procedure.
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (2) — Participant underwent surgical procedures for nasal obstruction at 519 and 682 days post procedure. Not related to the study device or procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-04): https://cdn.clinicaltrials.gov/large-docs/94/NCT03181594/Prot_SAP_000.pdf